CLINICAL TRIAL: NCT07008014
Title: What is the Scope for Low Field MRI to Replace Cone Beam Computed Tomography in Dentistry?
Brief Title: Can Dental Dedicated MRI Replace Low-dose CBCT Scanning in Dentistry
Acronym: DDMRI
Status: Not yet recruiting | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 328156; EDGE 166436 (Other: King's College London)
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-05

CONDITIONS: Dental Situations
Keywords: Dental; MRI
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients requiring orofacial imaging: Patients requiring orofacial imaging, provided their treating clinician would see significant value in obtaining an MRI image
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Participants will receive an additional MRI image in addition to standard of care to investigate if it was a useful imaging modality for their condition

SUMMARY:
Magnetic Resonance Imaging (MRI) has is a useful diagnostic tool that offers advantages over conventional radiography techniques. Unlike traditional X-ray or computed tomography (CT) scans, MRI utilizes a magnetic field and radio waves to generate detailed and high-resolution images of the body's internal structures. This non-invasive imaging modality allows the clinician to better see soft tissues in 3D without the use of ionising radiation. Furthermore, MRI enables the detection and characterization of a wide range of pathologies which can lead to improved diagnostic capabilities and better patient outcomes.

To date, the use of MRI in dentistry has been limited as dentistry imaging focuses predominantly on hard tissues (teeth and bones) in addition to the higher cost and accessibility issues with MRI machines.

However, recent developments have led to the development of a dental-specific coil for use with a low field strength (0.55 Tesla) MRI scanner. This has resulted in high diagnostic quality soft and hard tissue images and reduced imaging time. As this imaging modality has rarely been used before in dentistry, the aim of this study is to investigate its use for dental imaging, refining parameters and assessing the diagnostic quality of dental scans taken using MRI and the specific dental coil.

DETAILED DESCRIPTION:
The overall aim of this feasibility project is to optimise MRI parameters for dental use (i.e., dental-dedicated MRI) and assess the diagnostic quality of dental scans taken using MRI.

The objectives are to assess if MRI imaging has altered the diagnosis, retrospectively analyse the numbers of patients which can be diagnosed effectively using this radiation free imaging modality and document health resource use to inform a full health technology assessment trial.

The primary objective is to assess the feasibility of providing MRI scanning to dental patients and the resultant benefit. As such, the investigators will examine the percentage of patients whose diagnosis was altered as a result of additional MRI scanning.

The secondary objectives are to assess:

1. The percentage of patients who would have been able to complete their diagnosis with an MRI scan alone
2. Percentage of eligible patients who agreed to have an MRI scan
3. Percentage of patients who completed the MRI scan
4. Clinician rated diagnostic acceptability
5. Patient acceptability of the imaging modality (as determined by VAS scale)
6. Documentation of Health resource use including intervention costs

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 3 or over with suspected orofacial pathology involving a soft tissue component or healthy volunteers
2. The patient is willing to undergo an MRI investigation
3. Patient or their carer/guardian is able to provide informed consent to the study

Exclusion Criteria:

1. Patient or their carer is unable to show Gillick competency for consent.
2. The patient has pronounced claustrophobia.
3. The patient has a pacemaker or implanted defibrillator.
4. The patient has history of metal shrapnel injuries to the eyes or MRI incompatible metallic inclusions or implants/ large tattoos.
5. The patient has non-removable piercings.
6. Pregnant patients, or patients who suspect they could be pregnant
7. The patient has participated in other research studies within the previous 30 days.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients requiring orofacial imaging or healthy volunteers, provided their treating clinician would see significant value in obtaining an MRI image
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients whose diagnosis/care changed as a result of the additional dental MRI imaging compared to the total number of patients imaged using conventional radiography. | 4 weeks
  The treatment plan that was given before the MRI scan will be documented. Following review of the MRI by the overseeing consultant, any changes to the treatment plan will be documented. The number of patients whose treatment plan was altered as a result of the scan will be divided by the number of those who received a scan to get a percentage.
To assess diagnostic quality of the image | 6 months
  This is a feasibility trial and a new imaging modality for dentistry. Working with MR physicists we will assess image quality and report on areas for improvement

SECONDARY OUTCOMES:
Percentage of patients whereby the diagnosis could have been obtained using dental-dedicated MRI alone | 4 weeks
  The number of patients whereby the clinical indicators of pathology on the MRI scan were sufficient to gauge the pathology will be assessed. This will be divided by the number of patients who received a scan to get a percentage.
Time spent undergoing scan | 4 weeks
  Time spent undergoing scan (minutes)
Radiation exposure (Grays) | 4 weeks
  Radiation exposure of the imaging modality (Grays)

CONTACTS AND LOCATIONS:
Overall Officials: Saoirse O'Toole, BDentSc PhD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No
We can publish the results of the data but not participant scans or any identifiers.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT07008014/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT07008014/ICF_001.pdf